CLINICAL TRIAL: NCT01846403
Title: Feasibility and Acceptability of Using the Semi-quantitative Pregnancy Test to Replace Sequential Serum hCG Testing in an Assisted Fertility Setting
Brief Title: Feasibility and Acceptability of Using the Semi-quantitative Pregnancy Test in an Assisted Fertility Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6002
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semi-quantitative pregnancy test (Other): Semi-quantitative urine pregnancy test (dBest One Step hCG Panel Test Kit)
  Interventions: Device: Semi-quantitative urine pregnancy test

INTERVENTIONS:
Device: Semi-quantitative urine pregnancy test
  Other Names: (dBest One Step hCG Panel Test Kit)

SUMMARY:
Given the potential of semi-quantitative pregnancy tests as part of assisted fertility care, we would like to document the feasibility and acceptability of a semi-quantitative pregnancy test as an adjunct to or replacement of current monitoring protocols to offer women and health care providers a new choice of diagnostic tools to confirm early pregnancy. The pilot will help us to better understand how this tool complements existing monitoring protocols. If a suitable addition, replacement to repeat blood draws for serum hCG assessment, the SQPT could also contribute to efforts to make assisted fertility treatments more patient-friendly. This study seeks to test this innovation by asking women assigned to perform a dBest® semi-quantitative urine panel test (AmeriTekInc, Seattle WA, USA)at home on a weekly basis for up to 4 weeks after embryo transfer.

We hypothesize that the test, which can be used at home by women, will provide confirmation of the presence of a pregnancy compared with standard serum hCG testing because 1) it has sensitivity and specificity that correlates well with serum testing, and 2) it can be used at home and thus earlier to determine presence of hCG. Furthermore, a pregnancy can be assured only when a yolksac or embryo could be identified thus women have to wait for a period of 2-3 weeks after the next menses expected.

We hypothesize that women seeking assisted fertility treatments will be able to monitor their hCG at home as well. Further, we plan to develop revised instructions to better suit the needs and questions we think would be relevant to women desiring to use this test as part of assisted fertility services.

We hypothesize that the simple instructions we will develop for use in this study will enable women to use the test on their own. Provider counseling will complement these instructions and contribute to overall quality of care given to each participant.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for assisted fertility treatment according to hospital guidelines
* Agrees to have blood drawn several times for serum hCG tests
* Agrees to return for a series of follow-up visits
* Willing to follow provider instructions regarding use of at-home pregnancy test
* Willing to provide an address and/or telephone number to be contacted for purposes of follow-up
* Willing and able to consent to study participation

Exclusion Criteria:

* Women not eligible for assisted fertility treatment
* Women who do not agree to have blood drawn several times for serum hCG tests
* Women who do not agree return for a series of follow-up visits
* Women unable to follow provider instructions regarding use of at-home pregnancy test
* Women unable to provide contact information
* Women unable to sign the consent form

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Document whether continuing pregnancy can be successfully monitored at home using a semi-quantitative pregnancy test | 6 weeks

SECONDARY OUTCOMES:
Feasibility of women using this test at home on their own as a potential future substitute or complement to standard sequential clinic-based visits to monitor pregnancy after embryo transfer. | 6 weeks
Women's acceptability of using pregnancy tests at home instead of standard clinic-based monitoring after embryo transfer | 6 weeks
Assess if written instructions and provider's counseling enable women using the semi-quantitative pregnancy test at home to understand how it should be used and to correctly interpret the test result | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Thi Nhu Ngoc, MD, Principal Investigator — Center for Research and Consultancy in Reproductive Health; Ly Thai Loc, MD, Principal Investigator — Hungvuong Hospital; Tara Shochet, PhD, MPH, Principal Investigator — Gynuity Health Projects; Paul Blumenthal, MD, MPH, Principal Investigator — Stanford University; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (1):
- Hungvuong Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Shochet T, Comstock IA, Ngoc NTN, Westphal LM, Sheldon WR, Loc LT, Blum J, Winikoff B, Blumenthal PD. Results of a pilot study in the U.S. and Vietnam to assess the utility and acceptability of a multi-level pregnancy test (MLPT) for home monitoring of hCG trends after assisted reproduction. BMC Womens Health. 2017 Aug 22;17(1):67. doi: 10.1186/s12905-017-0422-y. PMID 28830483